CLINICAL TRIAL: NCT00325858
Title: Double-Blind, Randomized,Dose-Ranging, Parallel-Group Comparison Of The Efficacy And Safety Of Extended-Release Tramadol Hydrochloride(Tramadol HCl ER)100 Mg, 200 Mg, 300 Mg, And 400 Mg With Placebo In The Treatment Of Osteoarthritis Of Knee And/Or Hip
Brief Title: A Study Comparing the Effectiveness and Safety of Varying Dose Strengths (100, 200, 300 and 400 mg) of Extended-release Tramadol HCl With Placebo for the Treatment of Osteoarthritis(OA) of the Knee and/or Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B02.CT3.023.TRA P03
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2006-09

CONDITIONS: Chronic Pain
Keywords: osteoarthritis pain; knee; hip; extended-release analgesia; opioid
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tramadol HCl ER

SUMMARY:
The purpose of this study is to compare the effectiveness of multiple doses of once daily tramadol HCl ER (100, 200, 300 and 400 mg) to placebo in patients with moderate to severe pain due to OA. The study hypothesis is that tramadol HCl ER is safe and effective in the treatment of patients with moderate to severe pain due to OA.

DETAILED DESCRIPTION:
Immediate release (IR) tramadol has demonstrated efficacy in several pain conditions including: obstetrical, gynecological, orthopedic, abdominal, and oral surgery. The short elimination half-life of tramadol IR necessitates every 4-6 hour dosing to maintain optimal levels of analgesia in chronic pain. The study medication in this study is a once-daily, extended-release tramadol formulation. This is a 12-week multi-center, double-blind, randomized, dose-ranging, parallel-group, fixed-dose, placebo-controlled study. Patients with OA Functional Class I-III of the knee or hip (index joint) are eligible for participation, if appropriate criteria are met. During a 2-7 day washout period, the use of all analgesic medications will be discontinued. Eligible patients experiencing moderate to severe pain (<=40 mm on a 100 mm visual analog scale) in the index joint to be evaluated and who meet all other study criteria will enter in a 2-week,double-blind titration period. During this period, patients will be randomly assigned to receive treatment with tramadol HCl ER 100 mg, 200 mg, 300 mg, 400 mg or placebo, once a day. Patients will be titrated to their assigned dose between study days 1 - 15 and will continue at that dose for the remainder of the study (Week 12). Efficacy and safety evaluations will be collected at study visits occurring at Weeks 1, 2, 3, 6, 9 and 12 or at early termination. Study medication will be discontinued at Week 12 and patients will return after 1 week for a post-treatment visit (Week 13). Patients with unmanageable pain or with unacceptable side effects will be discontinued from the study and alternate analgesic therapy initiated, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American College of Rheumatology (ACR) Functional Class I-III OA of the knee or hip
* Patients with involvement of at least one knee or hip joint that warrants treatment with COX-2 inhibitors, NSAIDS, acetaminophen, or opioid analgesics for at least 75 of the 90 days preceding the screening visit
* Patients with a pain intensity score in index joint >=40 mm on the visual analog scale (VAS) at the baseline visit
* Patients who are able to discontinue acetaminophen, NSAIDS, COX-2 selective inhibitors, and other analgesics during the washout period and throughout the study
* Patients who are able to understand the study procedures and complete pain scales

Exclusion Criteria:

* Patients with a medical condition, other than OA, uncontrolled with treatment or any clinically significant condition that, in the investigator's opinion, precludes study participation or interferes with the assessment of chronic pain and other OA symptoms
* Patients with a diagnosis of inflammatory arthritis, gout, pseudo-gout or Paget's disease, that, in the investigator's opinion, interferes with the assessment of pain and other symptoms of OA
* Patients with a diagnosis of chronic pain syndrome
* Patients with an ACR or a clinical diagnosis of fibromyalgia
* Patients with a clinically significant form of joint disease or prior joint replacement surgery at the index joint
* Patients with an anticipated need for surgery or other invasive procedure in the index joint

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-01; Study Completion 2003-12

PRIMARY OUTCOMES:
The primary outcome is the change from baseline to Week 12 in the WOMAC OA Index pain and physical function subscale scores and the patient global assessment of disease activity.

SECONDARY OUTCOMES:
The secondary outcomes include: the change from baseline in the daily arthritis pain intensity scores from patient diaries; WOMAC OA stiffness subscale score, OA pain intensity VAS for index and non-index joints, and Chronic Pain Sleep Inventory scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Altoona Center for Clinical Research, Duncansville, Pennsylvania, United States

REFERENCES:
- [Background] Gana TJ, Pascual ML, Fleming RR, Schein JR, Janagap CC, Xiang J, Vorsanger GJ; 023 Study Group. Extended-release tramadol in the treatment of osteoarthritis: a multicenter, randomized, double-blind, placebo-controlled clinical trial. Curr Med Res Opin. 2006 Jul;22(7):1391-401. doi: 10.1185/030079906X115595. PMID 16834838